CLINICAL TRIAL: NCT04471012
Title: Impact of The Individual Counseling Program Using The Transtheoretical Model For Polycystic Ovary Syndrome Management Among University Students
Brief Title: The Transtheoretical Model For Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, dilek öcalan, Principal Investigator, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 205-84
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: transtheoretical model; individual counselling; university students
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual counselling program (Experimental): An individual counseling program that was based on TM and included motivational interview techniques was given to the experimental group which involved general information about the importance of weight control, healthy diet, and exercise.
  The experimental group was given a Benefits of Healthy Diet and Physical Activity in PCOS Training Booklet during their first counseling session.
  Interventions: Other: Individual counselling program
- Standard Care (No Intervention): The progress of the participants in the control group was tracked routinely without any specific implementation. At the end of the study, the control group was also given the same booklet.

INTERVENTIONS:
Other: Individual counselling program — An individual counseling program that was based on TM and included motivational interview techniques was given to the experimental group which involved general information about the importance of weight control, healthy diet, and exercise.
  Benefits of Healthy Diet and Physical Activity in PCOS Training Booklet was given during their first counseling session.
  Arms: Individual counselling program

SUMMARY:
The main objective of this study was to investigate the impact of individual counseling programs which has been designed from the Transtheoretical Model (TM) suggesting a healthy diet and physical activity for the students diagnosed with PCOS in the management of their syndrome. The data for the analysis was drawn from a sample of 854 students at first and a totally of 67 students were administered the scales. The control (N=33) and experimental groups (N=34) were formed based on a simple randomization technique.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation
* absence of sexual activity
* belonging to the age group of 19-24
* absence of chronic diseases
* absence of any physical disability and a lack of mental disorders.

Exclusion Criteria:

* being on medicine
* scores of above 18.5 and below 30 on the Body Mass Index (BMI)

Ages: 19 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Anthropometric Measurement | 1st month
  Anthropometric measurements that are frequently used to evaluate the nutritional status of the individuals are weight and height will be combined to report BMI in kg/m2.
Anthropometric Measurement Change | 3rd month
  Anthropometric measurements that are frequently used to evaluate the nutritional status of the individuals are weight and height will be combined to report BMI in kg/m2.
Anthropometric Measurement Change | 5th month
  Anthropometric measurements that are frequently used to evaluate the nutritional status of the individuals are weight and height will be combined to report BMI in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek OCALAN, PhD, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No